CLINICAL TRIAL: NCT02751346
Title: Persistent Postsurgical Pain (PPSP) Following Cystectomy: A Survey and Sensory Examination
Brief Title: Persistent Pain After Cystectomy for Bladder Cancer
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201509131
Record Dates: First submitted 2016-04-20; First posted 2016-04-26 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Pain; Surgery; Post Operative Pain
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Pain: Patients with pain identified through the survey will be invited to undergo sensory assessment by quantitative sensory testing (QST) around the surgical scar and a control area: Thermal (cold and heat) detection and pain thresholds; mechanical detection and pain threshold; dynamic mechanical allodynia; temporal summation (wind-up).
- Patients without Pain: Patients without pain age and gender matched to patients with pain identified through the survey will be invited to undergo sensory assessment by quantitative sensory testing (QST) around the surgical scar and a control area: Thermal (cold and heat) detection and pain thresholds; mechanical detection and pain threshold; dynamic mechanical allodynia; temporal summation (wind-up).

SUMMARY:
This single-center, cross-sectional survey and sensory examination is conducted to determine the prevalence, sensory characteristics and risk factors of PPSP in patients who underwent cystectomy at Washington University/Barnes-Jewish Hospital between 2009 and 2015. Based on data from other lower abdominal surgeries, the investigators hypothesize that 10-15% of patients undergoing cystectomy will develop PPSP.

DETAILED DESCRIPTION:
Currently, open radical cystectomy (ORC) with urinary diversion is the standard treatment for patient with muscle-invasive organ-confined bladder cancer. ORC involves the complete resection of local metastatic disease and reconstruction of a functional urinary tract. Additionally, minimally invasive laparoscopic surgery was shown to be safe alternative to open radical cystectomy. A total of 29,719 patients underwent a form of cystectomy in the United States between 2009 and 2011. Both cystectomy procedures require a midline incision on the pubic symphysis, and as with virtually any surgical incision, it produces tissue injury and inflammation, which result is acute post-operative pain.

Acute pain after surgery typically subsides with tissue healing; however, some patients go on to develop persistent post-surgical pain (PPSP). It is estimated that 21-52% of people who had underwent thoracotomy, 21.5-47.3% of women who had breast surgery, and 4.7%-18% of people who had underwent abdominal surgery developed PPSP. The incidence of the condition varies substantially by the type of surgical procedure, which is also an important factor affecting the mechanism of PPSP. For example, while thoracic surgeries result in predominantly neuropathic pain due to intraoperative nerve injury, in hysterectomies and knee replacement surgeries the mechanisms of PPSP seem to be predominantly inflammatory. However, no data are currently available on the prevalence or potential mechanisms of PPSP after cystectomy.

Understanding the prevalence, risk factors, and the potential mechanisms underlying PPSP after cystectomy will serve the basis for investigating approaches for risk stratification and prevention of PPSP in bladder cancer patients undergoing the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18;
* Cystectomy for bladder cancer performed at Washington University/Barnes-Jewish Hospital between Jan 1, 2009 and June 30, 2015.

Exclusion Criteria:

Surveys will not be sent if any of the following criteria exist:

* Patient is deceased or has moved out of the United States.
* Preoperative record indicates multiple surgeries in the abdominopelvic region.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Survey: 383 patients who have undergone cystectomy at Washington University/Barnes-Jewish Hospital.
  Sensory testing: Considering 25-30% 5-year mortality rate after cystectomy for bladder cancer, we expect 10-15 subjects with PPSP and 10-15 age and gender matched controls to participate in the sensory testing portion.
Sampling Method: Non-Probability Sample
Enrollment: 383 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Ratio of participants reporting PPSP at the time of survey. | between 3 months to 6 years post surgery
  Presence of PPSP will be determined based on presence of pain in the pelvic area at the time of survey.

SECONDARY OUTCOMES:
Comparison of sensory findings between patients with PPSP and patients without PPSP after cystectomy. This specific aim will be attained by performing Quantitative Sensory Testing (QST). | 1 to 3 months post survey completion

CONTACTS AND LOCATIONS:
Overall Officials: Simon Haroutounian, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaufman DS, Shipley WU, Feldman AS. Bladder cancer. Lancet. 2009 Jul 18;374(9685):239-49. doi: 10.1016/S0140-6736(09)60491-8. Epub 2009 Jun 10. PMID 19520422
- [Background] Tang K, Li H, Xia D, Hu Z, Zhuang Q, Liu J, Xu H, Ye Z. Laparoscopic versus open radical cystectomy in bladder cancer: a systematic review and meta-analysis of comparative studies. PLoS One. 2014 May 16;9(5):e95667. doi: 10.1371/journal.pone.0095667. eCollection 2014. PMID 24835573
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Haroutiunian S, Nikolajsen L, Finnerup NB, Jensen TS. The neuropathic component in persistent postsurgical pain: a systematic literature review. Pain. 2013 Jan;154(1):95-102. doi: 10.1016/j.pain.2012.09.010. PMID 23273105
- [Background] McNicol ED, Schumann R, Haroutounian S. A systematic review and meta-analysis of ketamine for the prevention of persistent post-surgical pain. Acta Anaesthesiol Scand. 2014 Nov;58(10):1199-213. doi: 10.1111/aas.12377. Epub 2014 Jul 25. PMID 25060512
- [Background] Andreae MH, Andreae DA. Regional anaesthesia to prevent chronic pain after surgery: a Cochrane systematic review and meta-analysis. Br J Anaesth. 2013 Nov;111(5):711-20. doi: 10.1093/bja/aet213. Epub 2013 Jun 28. PMID 23811426
- [Background] Treede RD, Jensen TS, Campbell JN, Cruccu G, Dostrovsky JO, Griffin JW, Hansson P, Hughes R, Nurmikko T, Serra J. Neuropathic pain: redefinition and a grading system for clinical and research purposes. Neurology. 2008 Apr 29;70(18):1630-5. doi: 10.1212/01.wnl.0000282763.29778.59. Epub 2007 Nov 14. PMID 18003941
- [Background] Fruhstorfer H, Lindblom U, Schmidt WC. Method for quantitative estimation of thermal thresholds in patients. J Neurol Neurosurg Psychiatry. 1976 Nov;39(11):1071-5. doi: 10.1136/jnnp.39.11.1071. PMID 188989
- [Background] Yarnitsky D, Sprecher E, Zaslansky R, Hemli JA. Heat pain thresholds: normative data and repeatability. Pain. 1995 Mar;60(3):329-32. doi: 10.1016/0304-3959(94)00132-x. PMID 7596629
- [Background] Baumgartner U, Magerl W, Klein T, Hopf HC, Treede RD. Neurogenic hyperalgesia versus painful hypoalgesia: two distinct mechanisms of neuropathic pain. Pain. 2002 Mar;96(1-2):141-51. doi: 10.1016/s0304-3959(01)00438-9. PMID 11932070
- [Background] Magerl W, Wilk SH, Treede RD. Secondary hyperalgesia and perceptual wind-up following intradermal injection of capsaicin in humans. Pain. 1998 Feb;74(2-3):257-68. doi: 10.1016/s0304-3959(97)00177-2. PMID 9520240
- [Background] Price DD, Hu JW, Dubner R, Gracely RH. Peripheral suppression of first pain and central summation of second pain evoked by noxious heat pulses. Pain. 1977 Feb;3(1):57-68. doi: 10.1016/0304-3959(77)90035-5. PMID 876667
- [Background] Brandsborg B, Dueholm M, Nikolajsen L, Kehlet H, Jensen TS. A prospective study of risk factors for pain persisting 4 months after hysterectomy. Clin J Pain. 2009 May;25(4):263-8. doi: 10.1097/AJP.0b013e31819655ca. PMID 19590472
- [Background] Aasvang EK, Kehlet H. Persistent sensory dysfunction in pain-free herniotomy. Acta Anaesthesiol Scand. 2010 Mar;54(3):291-8. doi: 10.1111/j.1399-6576.2009.02137.x. Epub 2009 Oct 15. PMID 19839945
- [Background] Brandsborg B, Dueholm M, Kehlet H, Jensen TS, Nikolajsen L. Mechanosensitivity before and after hysterectomy: a prospective study on the prediction of acute and chronic postoperative pain. Br J Anaesth. 2011 Dec;107(6):940-7. doi: 10.1093/bja/aer264. Epub 2011 Sep 2. PMID 21890662
- [Background] Gore JL, Litwin MS, Lai J, Yano EM, Madison R, Setodji C, Adams JL, Saigal CS; Urologic Diseases in America Project. Use of radical cystectomy for patients with invasive bladder cancer. J Natl Cancer Inst. 2010 Jun 2;102(11):802-11. doi: 10.1093/jnci/djq121. Epub 2010 Apr 16. PMID 20400716
- [Background] Wallace MS, Wallace AM, Lee J, Dobke MK. Pain after breast surgery: a survey of 282 women. Pain. 1996 Aug;66(2-3):195-205. doi: 10.1016/0304-3959(96)03064-3. PMID 8880841